CLINICAL TRIAL: NCT00316394
Title: Improving Preventive Service Delivery at Adult Complete Health Check-Ups: the Preventive Health Evidence-Based Recommendation Form (PERFORM) Cluster Randomized Controlled Trial
Brief Title: Improving Preventive Service Delivery at Adult Complete Health Check-Ups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 02-178
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2006-04

CONDITIONS: Preventive Health Care
Keywords: Preventive Health Care; Annual Health Check-up; Primary Care; Reminders

INTERVENTIONS:
Device: Preventive Care Checklist Form

SUMMARY:
To determine the effectiveness of a single checklist reminder form to improve the delivery of preventive health services at adult health check-ups in a family practice setting.

ELIGIBILITY:
Inclusion Criteria:

* Adults older than 21 years of age who had an complete health check-up completed at the clinic during the study period.

Exclusion Criteria:

* Charts were excluded if the patient was younger than 21, an investigator completed the assessment or the encounter was disease/illness specific.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-11; Study Completion 2003-03

PRIMARY OUTCOMES:
Rates and relative risks (RR) of the performance of 13 preventive health maneuvers at baseline and post-intervention and the percentage of up-to-date preventive health services delivered per patient were compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Vinita Dubey, MD MPH, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada